CLINICAL TRIAL: NCT06433362
Title: A Single Arm, Open Label, Multi-center Study of Mitoxantrone Hydrochloride Liposome With Cyclophosphamide, Vincristine, Etoposide and Prednisone (CMOEP) in Treatment-Naive Patients With Peripheral T-Cell Lymphoma
Brief Title: CMOEP in the Treatment of Untreated Peripheral T-cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DED-PTCL-K07
Record Dates: First submitted 2024-05-15; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Peripheral T Cell Lymphoma
Keywords: Untreated Peripheral T-cell Lymphoma; Mitoxantrone hydrochloride liposome
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CMOEP (Experimental): Mitoxantrone Hydrochloride Liposome with Cyclophosphamide, Vincristine, Etoposide and Prednisone
  Interventions: Drug: CMOEP

INTERVENTIONS:
Drug: CMOEP — Drug: Mitoxantrone hydrochloride liposome Mitoxantrone hydrochloride liposome (18 mg/m^2) on day 1, every 3 weeks; Drug: Cyclophosphamide Cyclophosphamide(750 mg/m^2) on day 1,every 3 weeks; Drug: Vincristine Vincristine (1.4mg/ m2，Max dose 2mg) will be administered by an intravenous injection on day 1(Or at the discretion of the investigator, use other vinblastine drugs with the same mechanism, such as vindesine 3 mg/m2, the maximum dose of 4mg),every 3 weeks; Drug: Etoposide Etoposide (60 mg/ m2) will be administered by an intravenous infusion on day 1-3,every 3 weeks;

SUMMARY:
This is a prospective, single arm, multicenter study to evaluate the safety and efficacy of CMOEP in patients with untreated peripheral T-cell lymphoma.

DETAILED DESCRIPTION:
This is a single-arm, open label, multi-center clinical study to evaluate the safety and efficacy of mitoxantrone hydrochloride liposome in combination with Cyclophosphamide, Vincristine, Etoposide and Prednisone(CMOEP) in patients with untreated Peripheral T-cell Lymphoma.Mitoxantrone hydrochloride liposome will be given on day 1 at dose of 18 mg/m2 and be combined with cyclophosphamide, vincristine, etoposide and prednisone.Each cycle consists of 21 days. A maximum of 6 cycles of therapy are planned.

ELIGIBILITY:
Inclusion Criteria:

* 1.Subjects fully understand and voluntarily participate in this study and sign informed consent.

  2. Age ≥18, ≤70years(for 65-70 years old, researchers need to comprehensively evaluate the physical fitness and tolerance of patients), no gender limitation.

  3. Expected survival ≥ 3 months. 4.Histologically confirmed diagnosis of Peripheral T-cell lymphoma： 1) Peripheral T-cell lymphoma unspecified (ptcl-NOS) 2) Angioimmunoblastic T-cell lymphoma (AITL) 3) Anaplastic large T-cell lymphoma (ALCL), ALK+ 4) Anaplastic large T-cell lymphoma (ALCL), ALK- 5) Other subtypes of PTCL that the investigator think can be included in the group.

  5.No previous treatment for PTCL, including chemotherapy, targeted therapy, immunotherapy, local radiotherapy for lymphoma (except for local radiotherapy to alleviate tumor related symptoms), surgical treatment.

  6.Subjects must have at least one evaluable or measurable lesion per lugano2014 criteria: for lymph node lesions, the length and diameter should be >1.5cm; For non-lymph node lesions, the length and diameter should be >1.0cm.

  7.Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-1. 8.The following baseline laboratory criteria are required: Absolute neutrophil count (ANC) ≥1.5×10^9/L, Platelet count (PLT) ≥75×10^9/L, Hemoglobin(HB)≥ 90 g/L(Restriction may be relaxed in patients with bone marrow involvement, Absolute neutrophil count (ANC) ≥1.0×10^9/L, Platelet count (PLT) ≥50×10^9/L, Hemoglobin(HB)≥ 75g/L).

  9.Total Serum creatinine (Scr) ≤1.5X upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5X ULN(For patients with liver invasion ≤5X ULN), bilirubin (TBIL)≤1.5X ULN(For patients with liver invasion ≤3X ULN ).

Exclusion Criteria:

* 1.Subjects with a history of prior antitumor therapy. 2.Hypersensitivity to any study drug or its components. 3.Uncontrolled systemic diseases (such as active infection, uncontrolled hypertension, diabetes, etc.) 4.Heart function and disease meet one of the following conditions:1）Long QTc syndrome or QTc interval >480 ms;2）Complete left bundle branch block, grade II or III atrioventricular block;3）Serious and uncontrolled arrhythmias requiring drug treatment;4）New York Heart Association grade ≥ II;5）Cardiac ejection fraction (LVEF)<50%;6）A history of myocardial infarction, unstable angina pectoris, severe unstable ventricular arrhythmia or any other arrhythmia requiring treatment, a history of clinically serious pericardial disease, or ECG evidence of acute ischemia or active conduction system abnormalities within 6 months before recruitment.

  5.Hepatitis B and hepatitis C active infection (defined as hepatitis B virus surface antigen positive and hepatitis B virus DNA higher than 1x10^3 copy/mL; hepatitis C virus RNA high than 1x10^3 copy/mL).

  6.Human immunodeficiency virus (HIV) infection (HIV antibody positive). 7.Patients with other malignant tumors, except for effectively controlled non melanoma skin basal cell carcinoma, breast/cervical carcinoma in situ and other tumor during the past 5 years.

  8.Patients with primary or secondary central nervous system (CNS) lymphoma or history of CNS lymphoma.

  9.Pregnant and lactating women and patients of childbearing age who are unwilling to take contraceptive measures.

  10.Unsuitable subjects for this study determined by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate (CRR) | 2 year
  Response is assessed according to the lugano criteria.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 2 year
  Response is assessed according to the lugano criteria.
Progression-Free-Survival (PFS) | 2 year
  From the date of the first dose of therapy is given until disease progression, death or last follow-up.
Overall survival (OS) | 2 year
  From the date of inclusion to date of death, irrespective of cause.
Safety and Tolerability | From the first day of medication to 28 days after the last dose
  The safety of the drug was evaluated by NCI-CTC AE 5.0 standard.Hematologic and non-hematologic toxicity.
Changes in cardiac safety indicators | 2 year
  such as LVEF% change from baseline, cardiac injury indicators, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Huilai Zhang, Study Director — Department of Lymphoma, Tianjin Medical University Cancer Institute and Hospital; Qingyuan Zhang, Study Director — The Second Affiliated Hospital of Harbin Medical University
Locations (1):
- Tianjin Cancer Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No